CLINICAL TRIAL: NCT06192160
Title: A Phase 2 Randomized, Adaptive, Dose-Ranging, Open-Label Trial of Novel Regimens for the Treatment of Pulmonary Tuberculosis
Brief Title: Trial of Novel Regimens for the Treatment of Pulmonary Tuberculosis
Acronym: RAD-TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: TB Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5409; DOH-27-032024-5399 (Other: South African National Clinical Trial Registry (SANCTR))
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid; Rifampin; Pyrazinamide; Ethambutol; bedaquiline; pretomanid; Linezolid; PNU-100480

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: Standard of Care (SOC) (Active Comparator): * Weeks 1-8: INH 300 mg, RIF 600 mg, PZA weight-based, EMB weight-based
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Pyrazinamide; Drug: Ethambutol
- Arm 2: Bedaquiline (BDQ), Pretomanid (Pa), and Linezolid (LZD) (Experimental): * Weeks 1-8: BDQ 400 mg for 2 weeks and then 200 mg for 6 weeks, Pa 200 mg, LZD 600 mg
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid
- Arm 3A: BDQ, Pa and TBI-223 (1200 mg) (Experimental): * Weeks 1-8: BDQ 400 mg for 2 weeks and then 200 mg for 6 weeks, Pa 200 mg, TBI-223 1200 mg
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Bedaquiline; Drug: Pretomanid; Drug: TBI-223
- Arm 3B: BDQ, Pa and TBI-223 (2400 mg) (Experimental): * Weeks 1-8: BDQ 400 mg for 2 weeks and then 200 mg for 6 weeks, Pa 200 mg, TBI-223 2400 mg
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Bedaquiline; Drug: Pretomanid; Drug: TBI-223
- Arm 4A: BDQ, Pa and Sutezolid (SZD) (800 mg) (Experimental): * Weeks 1-8: BDQ 400 mg for 2 weeks and then 200 mg for 6 weeks, Pa 200 mg, SZD 800 mg
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Bedaquiline; Drug: Pretomanid; Drug: Sutezolid
- Arm 4B: BDQ, Pa and SZD (1600 mg) (Experimental): * Weeks 1-8: BDQ 400 mg for 2 weeks and then 200 mg for 6 weeks, Pa 200 mg, SZD 1600 mg
  * Weeks 9-26: INH 300 mg, RIF 600 mg
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Bedaquiline; Drug: Pretomanid; Drug: Sutezolid

INTERVENTIONS:
Drug: Isoniazid — INH 300 mg will be administered as one tablet orally once daily.
  Other Names: INH
Drug: Rifampicin — RIF 600 mg will be administered as two 300 mg capsules orally once daily on an empty stomach, 1 hour before or 2 hours after eating a meal.
  Other Names: RIF
Drug: Pyrazinamide — PZA will be administered as 500 mg tablets, based on weight, orally once daily.
  Other Names: PZA
  Arms: Arm 1: Standard of Care (SOC)
Drug: Ethambutol — EMB will be administered as 400 mg tablets, based on weight, orally once daily.
  Other Names: EMB
  Arms: Arm 1: Standard of Care (SOC)
Drug: Bedaquiline — BDQ 400 mg will be administered as four 100 mg tablets orally once daily with a meal for the first 2 weeks followed by 200 mg (two 100 mg tablets) orally once daily with a meal for 6 weeks.
  Other Names: BDQ
  Arms: Arm 2: Bedaquiline (BDQ), Pretomanid (Pa), and Linezolid (LZD); Arm 3A: BDQ, Pa and TBI-223 (1200 mg); Arm 3B: BDQ, Pa and TBI-223 (2400 mg); Arm 4A: BDQ, Pa and Sutezolid (SZD) (800 mg); Arm 4B: BDQ, Pa and SZD (1600 mg)
Drug: Pretomanid — Pa 200 mg will be administered as one 200 mg tablet orally once daily with a meal.
  Other Names: Pa
  Arms: Arm 2: Bedaquiline (BDQ), Pretomanid (Pa), and Linezolid (LZD); Arm 3A: BDQ, Pa and TBI-223 (1200 mg); Arm 3B: BDQ, Pa and TBI-223 (2400 mg); Arm 4A: BDQ, Pa and Sutezolid (SZD) (800 mg); Arm 4B: BDQ, Pa and SZD (1600 mg)
Drug: Linezolid — LZD 600 mg will be administered as one 600 mg tablet orally once daily.
  Other Names: LZD
  Arms: Arm 2: Bedaquiline (BDQ), Pretomanid (Pa), and Linezolid (LZD)
Drug: TBI-223 — TBI-223 2400 mg once daily will be administered as four 600 mg tablets orally once daily with a meal.
  Arms: Arm 3B: BDQ, Pa and TBI-223 (2400 mg)
Drug: Sutezolid — SZD 1600 mg once daily will be administered as four 400 mg tablets orally once daily with a meal.
  Other Names: SZD
  Arms: Arm 4B: BDQ, Pa and SZD (1600 mg)
Drug: TBI-223 — TBI-223 1200 mg once daily will be administered as two 600 mg tablets orally with a meal.
  Arms: Arm 3A: BDQ, Pa and TBI-223 (1200 mg)
Drug: Sutezolid — SZD 800 mg once daily will be administered as two 400 mg tablets orally once daily with a meal.
  Other Names: SZD
  Arms: Arm 4A: BDQ, Pa and Sutezolid (SZD) (800 mg)

SUMMARY:
A5409/RAD-TB is an adaptive Phase 2 randomized, controlled, open-label, dose-ranging, platform protocol to evaluate the safety and efficacy of multidrug regimens for the treatment of adults with drug-susceptible pulmonary tuberculosis (TB).

A5409 hypothesizes that novel regimens for the treatment of pulmonary tuberculosis will result in superior early efficacy, as determined by longitudinal mycobacteria growth indicator tube (MGIT) liquid culture time to positivity (TTP) measurements over the first 6 weeks of treatment, and will have acceptable safety and tolerability over 8 weeks of treatment relative to standard of care [(SOC) isoniazid/rifampicin/pyrazinamide/ethambutol (HRZE)].

The study will run for 52 weeks, inclusive of 26 weeks of TB treatment comprised of 8 weeks of experimental or SOC treatment (based on treatment arm assignment) followed by 18 weeks of SOC treatment with 45 participants in each experimental treatment arm and at least 90 participants in the SOC arm.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary TB (among individuals either without history of prior TB treatment or with history of TB treatment more than 5 years prior to study entry), identified within 7 days prior to study entry by at least one sputum specimen positive for Mtb by Xpert. Semiquantitative Mtb results of "medium" or "high" are required.
2. Pulmonary TB with documented INH susceptibility (by Line Probe Assay (LPA) or Xpert MTB/XDR or other validated molecular test) and with documented RIF susceptibility (by LPA or Xpert MTB/RIF or Xpert MTB/RIF Ultra or other validated molecular test) within 7 days prior to study entry.
3. Documentation of HIV-1 infection status, as below:

   * Presence or Absence of HIV-1 infection, as documented by:

     * Any licensed rapid HIV test or HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit, any time prior to study entry. AND
   * Confirmed by one of the following:

     * A second antibody test from different manufacturers or based on different principles and epitopes (combination antigen-antibody-based rapid tests may be used), or
     * HIV-1 antigen, or
     * Plasma HIV-1 RNA viral load, or
     * A licensed Western blot
4. For individuals with HIV: CD4+ cell count ≥100 cells/mm3 based on testing performed within 30 days prior to study entry.
5. For individuals with HIV: Currently being treated with dolutegravir-based antiretroviral therapy (ART), or plan to initiate dolutegravir-based ART at or before study week 8.
6. Individuals age ≥18 years.
7. The following laboratory values obtained within 7 days prior to study entry at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs:

   * Serum or plasma alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN)
   * Serum or plasma total bilirubin ≤2 times ULN
   * Serum or plasma creatinine ≤2 times ULN
   * Serum or plasma potassium ≥3.5 mEq/L
   * Serum or plasma magnesium ≥1.0 mEq/L (≥0.500 mmol/L)
   * Absolute neutrophil count (ANC) ≥1500/mm^3
   * Hemoglobin ≥9.5 g/dL for individuals assigned to female sex at birth and ≥10.0 g/dL for individuals assigned to male sex at birth
   * Platelet count ≥100,000/mm^3
   * Negative for hepatitis B core antibody (HBcAb) total, hepatitis B surface antigen (HBsAg)
   * Negative for hepatitis C virus (HCV) antibody (or if HCV antibody positive, must have a negative HCV PCR)
8. For individuals assigned to female sex at birth and who are of reproductive potential, negative pregnancy test (urine HCG or serum β-HCG) within 3 days (72 hours) prior to entry by any network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

   Individuals assigned to female sex at birth, who are of reproductive potential, and who participate in sexual activity that could lead to pregnancy must agree to use at least two of the following forms of birth control while receiving TB study medications and for 12 months after stopping study medications:
   * Male or female condoms
   * Diaphragm or cervical cap (with spermicide, if available)
   * Intrauterine device (IUD) or intrauterine system (IUS)
   * Hormone-based birth control (e.g., oral contraceptives, Depo-Provera, NuvaRing, implants)
9. For individuals who are assigned male sex at birth who engage in sexual activity that may lead to pregnancy in their partner must agree to either remain abstinent or use male contraceptives. They are also strongly advised to inform their non-pregnant sexual partners of reproductive potential to use effective contraceptives while the individual is on study and for 90 days after experimental treatment discontinuation.
10. For individuals assigned male sex at birth with pregnant partners, willingness to use condoms during vaginal intercourse while on study and for 90 days after experimental treatment discontinuation.
11. For individuals assigned male sex at birth, willingness to refrain from sperm donation while on study and for 90 days after experimental treatment discontinuation.
12. Documentation of Karnofsky performance score ≥60 obtained within 14 days prior to study entry.
13. Chest x-ray obtained within 14 days prior to study entry.
14. A verifiable address or residence readily accessible for visiting, and willingness to inform the study team of any change of address during study treatment and follow-up period.
15. Ability and willingness of individual to provide informed consent.

Exclusion Criteria:

1. More than cumulative 7 days of treatment directed against active TB for the current TB episode in the 60 days preceding study entry.
2. Current extrapulmonary TB, in the opinion of the investigator.
3. QTcF interval >450 ms within 7 days prior to study entry.
4. History of or ongoing heart failure.
5. Personal or family history of congenital QT prolongation.
6. History of known, untreated, ongoing hypothyroidism.
7. History of or ongoing bradyarrhythmia.
8. History of torsades de pointes.
9. Current Grade 2 or higher peripheral neuropathy.
10. Other medical conditions (e.g., diabetes, liver or kidney disease, blood disorders, chronic diarrhea), in the opinion of the site investigator, in which the current clinical condition of the participant is likely to prejudice the response to, or assessment of, treatment.
11. Pregnant or breastfeeding or planning to become pregnant within the next 12 months.
12. Weight <35 kg.
13. Unable to take oral medications.
14. Taking any of prohibited medications.
15. Known allergy/sensitivity or any hypersensitivity to components of investigational agents or their formulation.
16. Active drug or alcohol use or dependence; or mental illness (e.g., major depression) that, in the opinion of the site investigator, would interfere with adherence to study requirements.
17. Taking an investigational drug or vaccine within 30 or more days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Difference in mean log10 (Time to positivity (TTP)) slope from longitudinal mycobacteria growth indicator tube (MGIT) liquid culture measurements over the first 6 weeks of treatment | Weeks 0, 1, 2, 3, 4 and 6
  for each experimental treatment arm compared to the SOC arm.
Difference in the cumulative proportion of participants having at least one new Grade 3 or higher adverse event (AE) by week 8 of treatment | 8 weeks
  for each experimental treatment arm compared to the SOC arm.

SECONDARY OUTCOMES:
Cumulative proportion of participants with stable sputum culture conversion by week 8 as measured by culture-negative status via MGIT liquid culture at two consecutive measurements. | 8 weeks
Mean log10 TTP slope from longitudinal MGIT liquid culture measurements over the first 8 weeks of treatment. | Weeks 0, 1, 2, 3, 4, 6 and 8
Cumulative proportion of participants with a new Grade 3 or higher AE by week 26 of treatment. | 26 weeks
Cumulative proportion of participants with permanent discontinuation of study-provided anti-TB drugs due to any reason prior to Week 8 of treatment. | 8 weeks
Cumulative proportion of participants with permanent discontinuation or temporary discontinuation for ≥3 days of at least one anti-TB drug due to any reason prior to week 8 of treatment. | 8 weeks
Cumulative proportion of participants with permanent discontinuation of at least one anti-TB drug due to any reason prior to week 26 of treatment. | 26 weeks
A composite of stable culture conversion at week 6 of treatment and no new Grade 3 or higher AE through week 8. | 8 weeks
Proportion of participants with durable cure by 52 weeks after treatment initiation. | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Radojka Savic, PharmD, PhD, Study Chair — University of California; Kelly Dooley, MD, PhD, Study Chair — Vanderbilt University Medical Center; Gustavo Velásquez, MD, MPH, Study Chair — University of California
Locations (28):
- 12701, Gaborone CRS, Gaborone, Botswana
- Brazil (2):
  - 12201, Hospital Nossa Senhora da Conceicao CRS, Porto Alegre
  - 12101, Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Haiti (2):
  - 30022, Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince
  - 31730, GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
- 31441, Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, India
- Kenya (2):
  - 12601, Moi University Clinical Research Center (MUCRC) CRS, Eldoret
  - 12501, Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho
- Malawi (2):
  - 30301, Blantyre CRS, Blantyre
  - 12001, Malawi CRS, Lilongwe
- 32078, Nutrición-Mexico CRS, Mexico City, Mexico
- Peru (2):
  - 11301, Barranco CRS, Lima
  - 31985, Socios En Salud Sucursal Perú CRS, Lima
- 31981, TB HIV Innovations and Clinical Research Foundation Corp., Cavite, Philippines
- South Africa (7):
  - 31793, South African Tuberculosis Vaccine Initiative (SATVI) CRS, Cape Town
  - 31792, University of Cape Town Lung Institute (UCTLI) CRS, Cape Town
  - 31422, CAPRISA eThekwini CRS, Durban
  - 11201, Durban International CRS, Durban
  - 12301, Soweto ACTG CRS, Johannesburg
  - 11101, University of the Witwatersrand Helen Joseph (WITS HJH) CRS, Johannesburg
  - 31684, Rustenburg CRS, Rustenburg
- Thailand (3):
  - 31784, Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
  - 5116 Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Rai
  - 31802, Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan
- Uganda (2):
  - 12401, Joint Clinical Research Centre (JCRC)/Kampala CRS, Kampala
  - 30293 MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala
- 32483 National Lung Hospital CRS, Hanoi, Vietnam
- 30313, Milton Park CRS, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Harrison LJ, Velasquez GE, Kempker RR, Imperial MZ, Nuermberger E, Dorman SE, Ignatius E, Granche J, Phillips PPJ, Furin J, Yang E, Foley C, Chiambah S, Rogers R, Van Grack A, Roa J, Shenje J, Nerette S, Kanyama C, Kyeyune RB, Mendoza-Ticona A, Murtaugh W, Foraida S, Goth M, Vernon A, Dooley KE, Savic RM. ACTG A5409 (RAD-TB): Study protocol for a phase 2 randomized, adaptive, dose-ranging, open-label trial of novel regimens for the treatment of pulmonary tuberculosis. Trials. 2025 Aug 15;26(1):291. doi: 10.1186/s13063-025-08973-w. PMID 40817073
- [Derived] Harrison L, Velasquez GE, Kempker RR, Imperial MZ, Nuermberger E, Dorman SE, Ignatius E, Granche J, Phillips PP, Furin J, Yang E, Foley C, Chiambah S, Rogers R, Van Grack A, Roa J, Shenje J, Nerette S, Kanyama C, Kyeyune RB, Mendoza-Ticona A, Murtaugh W, Foraida S, Goth M, Vernon A, Dooley KE, Savic RM. ACTG A5409 (RAD-TB): Study Protocol for a Phase 2 Randomized, Adaptive, Dose-Ranging, Open-Label Trial of Novel Regimens for the Treatment of Pulmonary Tuberculosis. Res Sq [Preprint]. 2025 Mar 26:rs.3.rs-5931694. doi: 10.21203/rs.3.rs-5931694/v1. PMID 40195983